CLINICAL TRIAL: NCT06654362
Title: The Effect of Multimodal Nutrition Intervention on Glucose and Lipid Parameters of Arfa Iron and Steel Company Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peyman Sarsangi (Other)
Responsible Party: Sponsor-Investigator, Peyman Sarsangi, Mr. Peyman Sarasangi, [Principal Investigator], Shahid Sadoughi University of Medical Sciences and Health Services
Organization: Shahid Sadoughi University of Medical Sciences and Health Services (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRSSU.SPHREC.1402.042
Record Dates: First submitted 2024-10-17; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Blood Sugar; Lipid Profile; Weight Change
Keywords: public health; workers; nutrition
MeSH Terms: conditions — Body Weight Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arfa's company workers (Experimental): all interventions administer to this arm
  Interventions: Behavioral: nutritional interventions include education and modifying company's restaurant menu

INTERVENTIONS:
Behavioral: nutritional interventions include education and modifying company's restaurant menu — * Reducing fried foods and replacing them with healthier alternatives.
  * Decreasing the consumption of sweetened beverages such as soda and replacing them with yogurt.
  * Reducing the intake of refined grains and substituting with whole grains.
  * Increasing fruit intake.
  * Increasing the intake of vegetables as much as possible.
  * Organizing face-to-face educational sessions with the chef to train them and improve cooking methods, to reduce fat and oil intake.

SUMMARY:
The goal of this clinical trial is to investigate the impact of nutritional interventions on glycemic and lipid profile factors among workers.

The main questions it aims to answer are:

Does nutritional interventions (include: nutritional education and Change in the Factory Restaurant's Menu improve glycemic and lipid profile factors among workers? Researchers will compare glycemic and lipid profile factors among workers before and after nutritional intervention .

ELIGIBILITY:
Inclusion Criteria:

* be Arfa's company worker

Exclusion Criteria:

* individuals who were diagnosed with any type of cancer

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1097 (Actual)
Dates: Start 2023-09-23 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Total Cholesterol, mg/dL | From enrollment to the end of intervention at 6 months
Total triglycerides, mg/dL | From enrollment to the end of intervention at 6 months
Low-density lipoprotein, mg/dL | From enrollment to the end of intervention at 6 months
High-density lipoprotein, mg/dl | From enrollment to the end of intervention at 6 months
Fast blood sugar, mg/dL | From enrollment to the end of intervention at 6 months
serum glutamic oxaloacetic transaminase, IU/L | From enrollment to the end of intervention at 6 months
serum glutamic pyruvic transaminase, IU/L | From enrollment to the end of intervention at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shahid Sadoughi University of Medical Sciences, Yazd, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarsangi P, NikAsa S, Ganji J, Fallahzadeh H, Nadjarzadeh A. The effect of multimodal nutrition intervention on glucose and lipid parameters of Arfa Iron and Steel Company workers. BMC Nutr. 2025 Jul 4;11(1):124. doi: 10.1186/s40795-025-01063-9. PMID 40615890